CLINICAL TRIAL: NCT05829265
Title: Non-randomised Feasibility Study Testing a Primary Care Intervention to Promote Engagement in an Online Health Community (OHC) for Adults With Troublesome Asthma
Brief Title: Feasibility of an Asthma Online Social Intervention
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); City, University of London (Other); University of Cambridge (Other); University of Edinburgh (Other); University of Nottingham (Other); University of Surrey (Other); St George's, University of London (Other); Asthma UK (Other)
Responsible Party: Sponsor
Other Study IDs: 314672
Record Dates: First submitted 2023-02-21; First posted 2023-04-25 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Asthma Intermittent, Uncontrolled

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group in the feasibility study.: There will only be one group in the feasibility study (i.e. all 50 patients recruited will receive the intervention).
  Interventions: Behavioral: A digital social intervention by primary care clinicians.

INTERVENTIONS:
Behavioral: A digital social intervention by primary care clinicians. — The intervention in this study will involve a structured consultation with a primary care clinician (e.g. a general practitioner (GP) or practice nurse) to promote online peer support, followed by engagement with the OHC of the Asthma + Lung UK (ALUK) charity. The intervention will either be delivered in person (in the general practices) or virtually. The aim is for the intervention to involve a face-to-face, one-off consultation, lasting approximately 30 minutes, during which a primary care clinician will:
  * Signpost and sign patients up to the ALUK OHC, by thoroughly explaining terms of conditions of use and providing log in details.
  * Introduce norms and values for passive (just reading) and active (writing OHC posts) participation.
  * Encourage seeking and offering self-management information and support, by emphasising that the OHC could be used ad hoc (e.g. when feeling unwell, or when there are information or emotional needs).

SUMMARY:
The goal of this observational study is to test the feasibility and acceptability of an online intervention for people with troublesome asthma in primary care, involving a consultation with a primary care clinician to introduce and promote online peer support (i.e. support from other patients with asthma within an established and safe OHC). The main questions this study aims to answer are:

* Is the intervention feasible and acceptable to patients?
* Can the research team recruit patients and collect health-related data to identify the impact of this intervention on patients and what are the challenges to pursue further research to evaluate this intervention in a trial?

DETAILED DESCRIPTION:
This observational study will involve a non-randomised, mixed-methods, feasibility study, setting out to test and refine a digital social intervention for people with troublesome asthma in primary care. The feasibility study will consist of a number of steps, including a questionnaire survey to identify and recruit eligible patients, intervention delivery, collection of follow-up outcomes, and exit one-to-one interviews with a sample of patients and primary care clinicians. Provided the feasibility study is successful, there are plans to undertake a full randomised controlled trial.

The precise content of the survey is currently being co-developed with stakeholders. However, the research team envisages including questions about participants' demographic and socioeconomic data, asthma symptoms, control and self-management, quality of life, mental wellbeing, health literacy, and interest in digital social interventions. Completion of the survey should take around 15 minutes.

Eligible patients identified through the survey will be invited to receive the intervention (see 'Groups and Interventions' section below). The exact content of the intervention is still being co-developed with patients and clinicians. Clinicians delivering the intervention will be thoroughly trained (through an online workshop/session) on the practicalities of signing patients up to an OHC, including on seeking and recording consent and collecting baseline data. The precise content of training is still being developed in collaboration with various stakeholders.

A number of outcomes, both self-reported and non-self-reported by patients, will be collected (see 'Outcome measures' section below). The self-reported outcome variables will be collected, via an online form designed on RedCap software, at baseline and at six months following the intervention. For the baseline collection, clinicians will add patients' responses to the online form at the time of delivering the intervention. For the follow-up collection, participants will receive a link to the online form, via a text message from the practice with which participants are registered, for self-submission (form completion should take 10-15 minutes).

A sample of patients and clinicians will be invited to participate in a one-to-one, semi-structured interview. Clinicians will be interviewed shortly after delivering the intervention to all recruited patients, whereas patients will be interviewed at the end of the feasibility study (i.e. after the completion of the follow-up period). An interview topic guide composed of open-ended questions and prompts will be used to elicit experiences of delivering/receiving the intervention. Based on individual participants' preferences, interviews will take place either in person (within private meeting or consultation spaces in the general practices) or virtually (via Zoom platform). Interviews should last approximately 30-90 minutes, depending on how much each participant has to share, and will be audio recorded through digital recorders or by using the Cloud function in Zoom. Basic demographic data will be collected at the time of the interview.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for receiving the intervention in the feasibility study:

* Patients with a diagnosis of asthma indicated in online clinical records.
* Aged 16 years and above.
* Have expressed, in the questionnaire survey, interest in receiving a digital social intervention.
* Experience troublesome asthma (i.e. asthma control test (ACT) score of less than 20).
* Sufficiently fluent in English to take part in a consultation and subsequent data collection procedures.
* Competent to consent for themselves, as determined by a qualified primary care healthcare professional.

Exclusion Criteria:

Patients who are

* Palliative or end-of-life.
* Receiving institutional long-term care (i.e. receiving total care in residential homes or living in nursing homes).
* Already a member of the ALUK OHC or other asthma OHCs/Facebook groups (general use of social media will not prevent participation).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three to six general practices in North and East London will act as recruitment sites. In each practice, a GP or nurse will create a list of all adults with a diagnosis of asthma, who are not receiving palliative/end of life or institutional care. These adults will receive a text message inviting them to take part in the online questionnaire survey. Patients fulfilling the inclusion criteria will be identified, via the survey, and invited to receive the intervention. Eligible patients will be purposively sampled so that a range of ethnic/age groups, health literacy levels, ACT score ranges and co-existing conditions are represented in the cohort of patients receiving the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients on the asthma register in the recruited practices | Baseline
  The number of patients on the asthma register will be measured in each recruited general practice, by extracting this information from practice records.
Number of: survey respondents, patients willing and unwilling to receive the intervention, participants who withdraw or have missing data | Through study completion, an average of 1 year
  Number of survey respondents and patients willing and unwilling to receive the intervention will be calculated from survey data, whereas number of participants who withdraw or have missing data will be obtained from the study's database.
Characteristics of: survey respondents, patients willing and unwilling to receive the intervention, participants who withdraw or have missing data | Through study completion, an average of 1 year
  Characteristics of survey respondents and patients willing and unwilling to receive the intervention will be obtained from survey data, whereas characteristics of participants who withdraw or have missing data will be obtained from the study's database.
Recruitment rate (i.e. proportion of asthma register and/or survey respondents interested in and eligible for the intervention) | Through study completion, an average of 1 year
  This proportion will be calculated based on the survey data and clinical records in the general practices used as recruitment sites.
Uptake rate (i.e. proportion of eligible patients consenting to the intervention and/or actively or passively engaging in the online health community (OHC) for the duration of the study) | Through study completion, an average of 1 year
  The proportion of patients consenting to the study will be calculated based on data from the survey and the study's database, whereas the proportion of patients engaging with the OHC will be calculated based on OHC activity data.
Retention rate (i.e. proportion of patients providing valid measures at the end of the follow-up period) | Through study completion, an average of 1 year
  This proportion will be based on data from the study's database.
Proportion of missing data (by outcome measure) | Through study completion, an average of 1 year
  This proportion will be based on data from the study's database.
Experience of patients receiving the intervention | Patient experiences will be obtained through study completion (an average of 1 year).
  Experiences of patients will be obtained via qualitative interviews with patients.
Experience of clinicians delivering the intervention | Clinician experiences will be obtained up to 24 weeks from study's commencement.
  Experiences of clinicians will be obtained via qualitative interviews with clinicians.

SECONDARY OUTCOMES:
Control of asthma | Baseline and at three months from intervention receipt.
  Control of asthma will be self-reported by patients through an Asthma Control Test (ACT) questionnaire.
Adherence to medications | Baseline and at three months from intervention receipt.
  Adherence to medications will be self-reported by patients through a MARS-10 questionnaire.
Number of asthma exacerbations over last 3 months | Baseline and at three months from intervention receipt.
  Asthma exacerbations will be self-reported by patients through a bespoke question.
Health-related quality of life | Baseline and at three months from intervention receipt.
  Health-related quality of life will be self-reported by patients through an EQ-5D-5L questionnaire.
Primary and secondary care use over last 3 months | Baseline and at three months from intervention receipt.
  Care use will be self-reported by patients through a bespoke question.
Time off work to seek care and/or due to asthma over last 3 months | Baseline and at three months from intervention receipt.
  Time off work will be self-reported by patients through a bespoke question.
Depression | Baseline and at three months from intervention receipt.
  Depression will be self-reported by patients through a PHQ-8 questionnaire.
Anxiety | Baseline and at three months from intervention receipt.
  Anxiety will be self-reported by patients through a GAD-7 questionnaire.
Self-efficacy | Baseline and at three months from intervention receipt.
  Self-efficacy will be self-reported by patients through the General Self-Efficacy Scale.
Amount of OHC engagement | Three months post intervention receipt.
  Amount of engagement with OHC will be self-reported by patients through a bespoke question.
Type (passive versus active) of OHC engagement | Three months post intervention receipt.
  Type of engagement with OHC will be self-reported by patients through a bespoke question.
Number of asthma exacerbations over last 3 months | Baseline and at three months from intervention receipt
  Exacerbations will be obtained from general practice records and data from the British Health Service (NHS)
Primary and secondary healthcare service utilisation over last 3 months | Baseline and at three months from intervention receipt
  Number of consultations in general practices, as well as number of hospital attendances and admissions, will be obtained from general practice records and data from NHS.
Costs associated with primary and secondary healthcare service utilisation over last 3 months | Baseline and at three months from intervention receipt
  Costs associated with primary care and hospital attendances, as obtained from general practice records and NHS data, will be calculated through economic models.
Amount of time spent on the OHC | Three months post intervention receipt
  Amount of time spent on the OHC will be provided to the research team by the manager of the ALUK OHC
Number of communities joined | Three months post intervention receipt
  Number of communities joined will be provided to the research team by the manager of the ALUK OHC
Number of logins to the OHC | Three months post intervention receipt
  Number of logins will be provided to the research team by the manager of the ALUK OHC
Number of likes on pages/posts within the OHC platform | Three months post intervention receipt
  Number of likes will be provided to the research team by the manager of the ALUK OHC
Time spent on pages within the OHC | Three months post intervention receipt
  Time spent on pages will be provided to the research team by the manager of the ALUK OHC
Public posts of the 50 participants within the OHC | Three months post intervention receipt
  Public posts will be provided to the research team by the manager of the ALUK OHC
Time of each public post in the OHC by the 50 participants | Three months post intervention receipt
  Time of posts will be provided to the research team by the manager of the ALUK OHC
Discussion thread of each public post in the OHC by the 50 participants | Three months post intervention receipt
  Discussion threads of each post will be provided to the research team by the manager of the ALUK OHC
User details in each discussion thread in the OHC in which one of the 50 participants was involved | Three months post intervention receipt
  User details in each discussion thread will be provided to the research team by the manager of the ALUK OHC
Time to deliver the intervention | Baseline
  This will be recorded by clinicians at the time of delivering the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anna De Simoni, PhD, Principal Investigator — Clinical Reader in Primary Care Research, Queen Mary University of London
Locations (1):
- CRN North Thames, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data from individual participants will not be shared. Participants will not be individually identifiable from any research outputs. 'Pseudonymisation of data' will be the policy for ensuring confidentiality. All participants will be coded, by allocating them unique participation codes. The association between participation codes and names will be contained on a Word/Excel document and will be stored on a password-protected computer at Queen Mary University of London. Any electronic documents or hard copies of data collected from participants will only be accessible to the research team. Only members of the research team will have access to associations between names and participation codes. Every attempt will be made to pool/aggregate or coarsely categorise potentially identifiable information in any dissemination of research findings.

REFERENCES:
- [Background] Karampatakis GD, Wood HE, Griffiths CJ, Taylor SJC, Toffolutti V, Bird VJ, Lea NC, Ashcroft RE, Day B, Coulson NS, Panzarasa P, Li X, Sheikh A, Relton C, Sastry N, Watson JS, Marsh V, Mant J, Mihaylova B, Walker N, De Simoni A. Non-randomised feasibility study testing a primary care intervention to promote engagement in an online health community for adults with troublesome asthma: protocol. BMJ Open. 2023 Jul 11;13(7):e073503. doi: 10.1136/bmjopen-2023-073503. PMID 37433727
- [Background] Karampatakis GD, Wood HE, Griffiths CJ, Lea NC, Ashcroft RE, Day B, Walker N, Coulson NS, De Simoni A. Ethical and Information Governance Considerations for Promoting Digital Social Interventions in Primary Care. J Med Internet Res. 2023 Sep 27;25:e44886. doi: 10.2196/44886. PMID 37756051